CLINICAL TRIAL: NCT00548743
Title: Practice Based Clinical Trial of Screening, Diagnosis and Follow up Management for Postpartum Depression in Family Medicine Practices.
Brief Title: Translating Research Into Practice for Postpartum Depression
Acronym: TRIPPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Olmsted Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 5R01HS014744-02 (AHRQ)
Record Dates: First submitted 2007-10-22; First posted 2007-10-24 (Estimated); Last update posted 2007-12-04 (Estimated); Status verified 2007-10

CONDITIONS: Postpartum Depression
Keywords: Depression; Postpartum; Dyad satisfaction; Parenting comfort; Screening; Management; Follow up; Primary care; Practice based research
MeSH Terms: conditions — Depression, Postpartum; Depression | interventions — Mass Screening

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Intervention arm
  Interventions: Behavioral: Screening and follow up
- 2 (Placebo Comparator): Usual care
  Interventions: Behavioral: Usual care

INTERVENTIONS:
Behavioral: Screening and follow up — Two stage screening with EPDS and PHQ-9, treatment for depression at physician's discretion and follow up phone calls and visits
  Arms: 1
Behavioral: Usual care — usual care for identification and management of postpartum depression
  Arms: 2

SUMMARY:
This is a study to assess the impact of introducing screening and planned follow up for postpartum depression. All women ages 18 to 45 who speak English or Spanish who come to the enrolled community family medicine offices will either be given usual care or screened using the Edinburgh Postnatal Depression Screening tool. If the EDPS score is high the women will be given the PHQ-9 to more clearly identify the specific likelihood of being depressed. Women who are determined to be depressed will be treated with medication or counseling based on the preference of the women and their physicians. Women will be followed through nurse initiated phone calls and visits to the physicians office.

Outcomes include the level of depression symptoms, measure of comfort with parenting, and satisfaction with partner relationships comparing baseline levels with those at 6 and 12 months from the usual care and intervention sites. These data will be collected by questionnaire. In addition, with the women's permission, medical records will be reviewed.

DETAILED DESCRIPTION:
A randomized controlled trial of screening and management of postpartum depression that includes a second phase assessing the maintenance of the intervention in the original intervention sites and a switch from usual care to intervention in the control sites.

Planned enrollment includes 29 family medicine practices and 3000 women over a period of four years. All follow up and management is initiated within the family medicine practices to improve generalizability and likelihood for dissemination.

In addition to the patient centered outcomes, exploratory analyses will look at the uptake and degree of implementation and maintenance of the intervention based on characteristics of the practice including size, location, affiliation with larger group, type of practice and whether or not the practice is a community health center or residency practice.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 12 weeks postpartum
* Able to speak and read English or Spanish

  * 18 to 45 years of age

Exclusion Criteria:

* Significant cognitive impairment and unable to answer screening questions

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3000 (Estimated)
Dates: Start 2005-09; Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Level of depressive symptoms and level of parenting comfort | 12 months postpartum

SECONDARY OUTCOMES:
Percent eligible women screened and of those screen positive, percent treated and followed according to protocol | 12 months for each women

CONTACTS AND LOCATIONS:
Overall Officials: Barbara P Yawn, MD MSc, Principal Investigator — Olmsted Medical Center
Locations (1):
- Olmsted Medical Center, Rochester, Minnesota, United States